CLINICAL TRIAL: NCT02097264
Title: A Randomised, Active Comparator, Double-blind, Multi Centre, Parallel, Phase 2a Trial, Investigating the Mechanism of Action, of NNC0109-0012 (Anti-IL-20 mAb) Through Synovial Biopsies in Subjects With Rheumatoid Arthritis and an Inadequate Response to Methotrexate
Brief Title: A Trial Investigating the Mechanism of Action of NNC0109-0012 (Anti-IL-20 mAb) Through Synovial Biopsies in Subjects With Rheumatoid Arthritis and an Inadequate Response to Methotrexate
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8226-4064; 2013-001492-20 (EudraCT Number); U1111-1141-3512 (Other: WHO); REec-2014-0740 (Registry Identifier: Spanish Register of Clinical Studies (REec))
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Inflammation; Rheumatoid Arthritis
MeSH Terms: conditions — Inflammation; Arthritis, Rheumatoid | interventions — Fletikumab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC0109-0012 (Experimental)
  Interventions: Drug: NNC0109-0012; Drug: placebo
- Adalimumab (Active Comparator)
  Interventions: Drug: Adalimumab; Drug: placebo

INTERVENTIONS:
Drug: NNC0109-0012 — Solution for injection administered subcutaneously (s.c. - under the skin). 240 mg NNC0109-0012 will be administered weekly for 12 weeks
  Arms: NNC0109-0012
Drug: Adalimumab — Solution for injection administered subcutaneously (s.c. - under the skin). Administered every other week for 12 weeks; Each active treatment involves 1 (one) s.c. injection of adalimumab 40 mg/0,8 mL solution for injection for paediatric use (Humira®)
  Arms: Adalimumab
Drug: placebo — Solution for injection administered subcutaneously (s.c. - under the skin).
  1 active adalimumab injection and 2 placebo injections per active treatment (every other week), and 3 placebo injections on placebo visits (alternative weeks).

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the mechanism of action of NNC0109-0012 (anti-IL-20 mAb) through synovial biopsies in subjects with rheumatoid arthritis (RA) and an inadequate response to Methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age at least 18 and below or equal to 75 years at the time of signing informed consent
* A diagnosis of RA at least 6 months prior to screening visit, according to the American College of Rheumatology (EULAR/ACR 2010 criteria) or by standard criteria (ACR 1987) if diagnosis was made earlier than 2010
* Subjects with ACR global functional status of 1 to 3
* Active RA, characterised by: DAS28 (Disease Activity Score 28) (CRP (C-reactive protein)) above 4.5 and equal to or above 6 tender and equal to or above 6 swollen joints based on a 66/68 joint count
* Active Synovitis in at least two joints of the wrist and metacarpophalangeal joints, as assessed by high frequency Power Doppler ultrasound scan at screening and randomisation

Exclusion Criteria:

* Subjects with arthritis due to other autoimmune diseases than RA
* Body weight above 90.0 kg
* History of or current inflammatory joint disease other than RA (e.g. gout, psoriatic or reactive arthritis, Lyme disease, juvenile idiopathic arthritis, excluding secondary Sjogren syndrome and hypothyroidism)
* Any active or on-going bacterial infections within 4 weeks prior to screening visit, unless treated and resolved with appropriate therapy or any history of recurrent infections or conditions predisposing to chronic infections (e.g., bronchiectasis, chronic osteomyelitis)
* Subjects with malignancy within the previous 5 years with the exception of adequately treated and cured basal or squamous cell carcinoma of the skin or cervical carcinoma in situ occurring more than 12 months prior to screening visit
* Female who is pregnant, breast feeding, intends to become pregnant or is of childbearing potential, not willing to use two highly effective contraceptive methods (adequate highlyeffective contraceptive measures are defined as established use of oral, injected or implanted hormonal methods of contraception, sterilisation, intrauterine device or intrauterine system) one of which has to be a barrier method a barrier method of contraception (e.g. condom with spermicidal foam/gel/film/cream), for at least 16 weeks (approximately 5 half-lives) following the last dose of trial medication
* Male subjects who are sexually active and not surgically sterilised, who or whose partner are unwilling to use two different forms of highly effective contraception, one of which has to be a barrier method a barrier method of contraception (e.g. condom with spermicidal foam/gel/film/cream) for the duration of the trial and for at least 16 weeks (approximately 5 half-lives) following the last dose of trial medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change in the total histopathological synovitis score | Week 0, week 12

SECONDARY OUTCOMES:
Change in dynamic contrast enhanced MRI (DCE-MRI) measures of initial rate of enhancement (IRE) | Week 0, week 12
Change in dynamic contrast enhanced MRI (DCE-MRI) measures of maximal enhancement (ME) | Week 0, week 12
Changes in RA-MRI scores (RAMRIS (Rheumatoid arthritis magnetic resonance imaging)) of synovitis | Week 0, week 12
Changes in RA-MRI scores (RAMRIS) of oedema | Week 0, week 12
Changes in RA-MRI scores (RAMRIS) of erosion | Week 0, week 12
Change in high frequency ultrasound with Power Doppler measures of total synovitis | Week 0, week 12
Change in high frequency ultrasound with Power Doppler measures of total tenosynovitis scores | Week 0, week 12
Change in disease activity 28 - C-reactive protein (DAS28 (CRP) | Week 0, week 12
Incidence of Adverse Events (AE) | Week 0, week 24
Incidence of local intolerability at the injection site | Week 0, week 24

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com